CLINICAL TRIAL: NCT04399499
Title: Use of Percutaneous Mitral Leaflet Approach for Severe Mitral Regurgitation in Cardiogenic Shock: Results From a Multicenter Observational Italian Experience (the Mitra-Shock Study).
Brief Title: Percutaneous Mitral Valve Repair in Cardiogenic Shock: Mitra-Shock Study
Acronym: MSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Agricola Eustachio, Professor, IRCCS San Raffaele
Other Study IDs: MITRA-SHOCK-2020
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Mitral Regurgitation Functional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: MitraClip implantation — The MitraClip® procedure is performed under general anesthesia and orotracheal intubation. The procedure is usually guided by 2 and 3-dimensional transesophageal echocardiography and fluoroscopy. This catheter-based technology is inserted through femoral venous access and advanced in the left atrium through the transseptal puncture. The MitraClip® is provided by 2 arms able to grasp the anterior and posterior mitral leaflets. The goal is to approximate both leaflets creating a double orifice mitral valve mimicking the edge-to-edge surgical repair procedure (Alfieri stitch).

SUMMARY:
Cardiogenic shock (CS) is a medical emergency and a frequent cause of death. CS can be complicated and/or precipitated by mitral regurgitation (MR). The efficacy of percutaneous treatment of MR in patients with cardiogenic shock is unknown. The aims of the study will be to analyse the efficacy of MitraClip therapy on early (30 days) and midterm mortality (6 months) as well as the predictors of outcomes. Investigators will also report the rate of periprocedural complications such as minor and major bleeding, vessel injury and Acute Kidney Injury (AKI).

It is a multicenter retrospective observational study on CE marked medical device (MitraClip® System). Retrospective time range: from 01/01/2012 to 01/01/2020

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old

Exclusion Criteria:

* multiorgan failure,
* VA-ECMO,
* inadequate peripheral access because of vascular disease,
* not suitable mitral valve anatomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CS and concomitant severe MR who underwent PMVR between 01/01/2012 to 01/01/2020 will be included in the study. Five Italian centers with high volume of MitraClip procedures will participate in the study. The number of enrolled patients will be of 30 patients. All patients will be older than 18 years old. Patients enrolled at our center (OSR) will be of 10 patients. The patients can tolerate antiplatelets and anticoagulant therapy. Inclusion criteria are: cardiogenic shock, severe mitral regurgitation, prohibitive surgical risk (STS>10%), anatomic feasibility of PMVR with MitraClip® system. Exclusion criteria are: multiorgan failure, VA-ECMO, inadequate peripheral access because of vascular disease, not suitable mitral valve anatomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
Mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided